CLINICAL TRIAL: NCT06589375
Title: Neuroscent: EEG Analysis of Cortical Signals Induced by Olfactory Stimuli in Normosmic Subjects and Individuals With Olfactory Disorders, With an In-depth Study of Olfactory Pathways in Patients With Tinnitus
Brief Title: Study of EEG and Nasal Stimulus in Olfactory Disorders
Acronym: SENSO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ID6911
Record Dates: First submitted 2024-08-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Olfaction Disorders
Keywords: Olfactory stimuli; EEG; Tinnitus; Olfactory disorders; Smell impairment; Olfactometry; Brain waves
MeSH Terms: conditions — Olfaction Disorders; Tinnitus | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: This study involves multiple groups of participants who will undergo EEG analysis during olfactory stimulation to assess brain wave responses. The groups include normosmics, hyposmics, tinnitus patients with hyposmia, and tinnitus patients without hyposmia. The study aims to differentiate between these groups and investigate the relationship between olfactory disorders and also highlight the olfactory features of patients with tinnitus. Each group will receive the same olfactory tests and EEG recordings, but they will be compared against each other to understand the different responses and interactions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normosmic (Active Comparator): Participants in this group have normal olfactory function, as determined by the Sniffin' Sticks test. They will undergo EEG analysis while being exposed to various olfactory stimuli to establish baseline brain wave patterns for normal olfactory responses.
  (n=550)
  Interventions: Diagnostic Test: Sniffin'Sticks
- Hyposmic (Active Comparator): Participants in this group have impaired olfactory function (hyposmia), confirmed through the Sniffin' Sticks test. They will undergo EEG analysis during olfactory stimulation to identify differences in brain wave patterns compared to normosmic individuals. (n=150)
  Interventions: Diagnostic Test: Sniffin'Sticks
- Tinnitus Patients with Hyposmia (Active Comparator): This group includes participants who have both tinnitus and hyposmia. They will be subjected to EEG analysis during olfactory testing to investigate the interaction between olfactory and auditory disorders and how these conditions may influence brain wave responses. (n=150)
  Interventions: Diagnostic Test: Sniffin'Sticks
- Tinnitus Patients without Hyposmia (Active Comparator): Participants in this group have tinnitus but normal olfactory function. They will undergo the same EEG and olfactory tests to explore the impact of tinnitus on brain wave patterns in the absence of olfactory disorders and to compare their responses with those of other groups. (n=150)
  Interventions: Diagnostic Test: Sniffin'Sticks

INTERVENTIONS:
Diagnostic Test: Sniffin'Sticks — The Sniffin' Sticks test, a validated method to evaluate olfactory functions, utilizes pen-like devices to dispense scents for testing identification, discrimination, and detection of odors. In this study, participants' responses to various scents are recorded. EEG (Electroencephalography) captures electrical activity in the brain during exposure to these odors by using an EEG cap fitted with electrodes on the scalp. This allows for the monitoring of brain wave patterns in response to olfactory stimuli. Both the Sniffin' Sticks test and EEG recordings are conducted simultaneously, providing a dual assessment of behavioral reactions and brain activity to odors. The goal of the study is to compare brain wave patterns and olfactory function in normosmic (normal smell), hyposmic (reduced smell), and tinnitus patients with and without olfactory impairments, delivering comprehensive insights into the neural basis of olfactory perception.
  Other Names: EEG

SUMMARY:
Neuroscent aims to analyze EEG signals induced by olfactory stimuli in individuals with normal and impaired olfactory functions, with a focus on patients with tinnitus. The study seeks to develop reliable diagnostic methods using EEG to differentiate between normosmic and hyposmic subjects during olfactory tests, potentially enhancing our understanding of the brain's response to olfactory stimuli. This 24-month interventional study with a device to be patented will involve 1000 participants and aims to establish more effective diagnostic and therapeutic tools for olfactory disorders

DETAILED DESCRIPTION:
The Neuroscent project investigates the EEG signals elicited by olfactory stimuli in both normosmic individuals and those with olfactory disorders, with a focus on tinnitus patients. The primary objective is to utilize EEG analysis to identify and quantify brain wave responses during olfactory tests with Sniffin' Sticks, aiming to accurately differentiate between normosmic and hyposmic subjects. This research aims to enhance the diagnostic precision and understanding of the interplay between olfactory and auditory stimuli in the brain. The 24-month, interventional study with a device to be patented, co-financed by the Ministry of Health and Ministry of the Interior under the PNRR 2023, will recruit 1000 participants divided into four groups: normosmics (550), hyposmics (150), tinnitus patients with hyposmia (150), and tinnitus patients without hyposmia (150). Participants will undergo comprehensive olfactory assessments, including the Sniffin' Sticks test, and EEG recordings will be taken during olfactory stimulation to capture brain wave patterns. Advanced data analysis techniques, such as Random Forest algorithms and t-SNE dimensionality reduction, will be employed to classify and interpret the EEG signals, aiming to develop effective diagnostic and therapeutic tools for olfactory disorders, thereby improving clinical outcomes and quality of life for affected individuals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age who have given consent for the collection of specified data, including medical history and personal information, for the purposes of project implementation and in accordance with the ethical standards of the institutions where the project will be conducted.

Exclusion Criteria:

* Previous fractures of the facial bones, particularly the ethmoid bone.
* Active tumors of the brain or face, including tumors of the nose, paranasal sinuses, oral cavity, or nasopharynx.
* Active nasal-sinus conditions, particularly radiologically proven sinusitis.
* Mass in the pontocerebellar angle, especially schwannoma of the VIII nerve.
* Patients with acute and chronic inflammatory diseases of the middle ear, otosclerosis, inner ear diseases (especially Meniere's disease), objective tinnitus, and tinnitus caused by middle ear pathologies and CPA tumors.
* Neurodegenerative diseases (especially Alzheimer's and Parkinson's disease).
* Known history of neuropsychiatric or cerebral disorders.
* Use of psychotropic drugs or drugs active on the central nervous system.
* Alcohol and drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment and data collection | 22 months
  During this period, 1000 participants > 18 y/o will be recruited and divided into four distinct groups: normosmics (550), hyposmics (150), tinnitus patients with hyposmia (150), and tinnitus patients without hyposmia (150). The primary outcome of the Neuroscent project is to assess the ability of EEG analysis to distinguish between normosmic and hyposmic participants during olfactory stimulation using the Sniffin' Sticks test.
EEG Parameters (in µV²) | 22 months
  Alpha Power: Measured in microvolts squared (µV²), representing the magnitude of Alpha wave activity during olfactory stimulation. Theta Power: Measured in microvolts squared (µV²), representing the magnitude of Theta wave activity during olfactory stimulation. We will make use of the Fourier transform as well, which is inherently dimensionless. The data acquisition setup involves placing blindfolded participants in an isolated room and administering three randomized olfactory stimuli (pure olfactory, trigeminal, and olfactory-gustatory) while collecting EEG data. Sessions start and end with a 30-second resting state.
Behavioral/Performance Measures (Scores) | 22 months
  Olfactory Threshold Scores (as per routinary diagnosis of olfactory performances): Derived from the Sniffin' Sticks test, these scores quantify participants' ability to detect odors, classifying them as normosmic or hyposmic. All the participants will undergo a complete olfactory assessment through the Sniffin' Sticks test. These are represented as numerical scores. The maximum score obtainable in the full Sniffin' Sticks test, which includes the three sub-tests (Threshold, Discrimination, Identification - TDI), is 48. This maximum score is achieved by summing the highest possible score from each of the three components: 16 for olfactory threshold (Threshold), 16 for olfactory discrimination (Discrimination), and 16 for olfactory identification (Identification).
Model Performance Metrics (Accuracy) | 22 months
  Random Forest Model Classification Accuracy: The accuracy of the classification model used to distinguish between normosmic and hyposmic participants based on EEG data, usually expressed as a percentage or a value between 0 and 1.
Dimensionality Change Outputs (t-SNE) | 22 months
  t-SNE Features: Although these don't have a specific unit, they represent the reduced dimensional data points used as features in the Random Forest model. These are typically dimensionless and used in the context of visualizing and improving model performance.

SECONDARY OUTCOMES:
Pure Tone Audiometry Test | 22 months (Simultaneously with the primary outcome)
  Pure Tone Audiometry (PTA), as per routinary diagnosis of Tinnitus: Measures hearing thresholds across frequencies, reported in decibels Hearing Level (dB HL) to determine the degree of hearing loss. The results are plotted on an audiogram, which shows the person's hearing threshold at different frequencies; a normal audiogram threshold is 0-20 dB HL between 250 and 8k Hz.
Behavioral/Performance Measures (Scores) | 22 months (Simultaneously with the primary outcome)
  Tinnitus Handicap Inventory (THI): Scores the impact of tinnitus on a scale from 0 to 100, where a higher score indicates a worse impact of tinnitus.
EEG Parameters | 22 months (Simultaneously with the primary outcome)
  EEG Data: Analyzed during exposure to olfactory stimuli (as per Primary Outcome), with features reduced via t-SNE and classified using a Random Forest algorithm.
Model Performance Metrics | 22 months (Simultaneously with the primary outcome)
  Random Forest Model Classification Accuracy: Measures the accuracy of the model used to classify participants across the four groups. This is typically expressed as a percentage or a value between 0 and 1. Fleiss' Kappa Statistic: Used to evaluate the agreement of classification, reported as a kappa coefficient.
Power Analysis and Post-hoc Analyses | 22 months (Simultaneously with the primary outcome)
  Power Analysis: Ensures the sample size is adequate to detect significant effects. This is typically expressed in terms of statistical power (e.g., 0.8 or 80%). Post-hoc Analyses: Conducted if significant differences are found, usually involving p-values or effect sizes.
Auditory Brainstem Response (ABR) | 22 months (Simultaneously with the primary outcome)
  Auditory Brainstem Response (ABR) as per routinary diagnosis of Tinnitus: Assesses the auditory nerve and brainstem's response to sound stimuli by measuring electrical activity in the brain. Results are typically presented as waveforms, with particular focus on latency and amplitude of specific waves, measured in milliseconds (ms) and microvolts (µV) respectively, to evaluate neural pathways involved in hearing.
Tympanometry | 22 months (Simultaneously with the primary outcome)
  Tympanometry, as per routinary diagnosis of Tinnitus: Evaluates middle ear function by measuring tympanic membrane mobility, with results reported in decapascals (daPa) and milliliters (mL). The pressure reading in tympanometry reflects the air pressure in the middle ear cavity. A normal tympanogram shows peak compliance when the pressure in the ear canal matches the pressure in the middle ear, indicating normal middle ear function. The two units of measurement, pressure and compliance, are plotted on a two-dimensional graph. Pressure (daPa) is plotted on the x-axis and compliance, measured in mL, is plotted on the y-axis in the two-dimensional graph

OTHER OUTCOMES:
Predicting Odor Categories in Tinnitus and Non-Tinnitus Groups Using EEG and Machine Learning | 2 months
  The final outcome will involve comparing olfactory perception across four participant groups (normosmic, normosmic with tinnitus, hyposmic, and hyposmic with tinnitus) using EEG features derived from Fourier analysis, reduced via t-SNE, and classified with a Random Forest algorithm. The model's accuracy in predicting odor categories (based on EEG data) will be evaluated using metrics such as accuracy, precision, recall, specificity, and F1 score. Fleiss' kappa statistic will assess agreement across groups, comparing the algorithm's predictions with the Sniffin' Sticks test results. Statistical power analysis ensures adequate sample sizes for reliable comparisons, with post-hoc analyses conducted if significant differences are detected.

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Cesare Passali, Prof, Study Director — Fondazione Policlinico Universitario A. Gemelli, IRCCS

IPD SHARING:
Plan to Share IPD: No